CLINICAL TRIAL: NCT05345678
Title: An Early Access Program for Durvalumab and Tremelimumab as First Line Treatment for Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Himalaya Early Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419CR00019
Record Dates: First submitted 2022-02-03; First posted 2022-04-26 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — durvalumab; tremelimumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Durvalumab — Dose: 1500mg Route: IV
  Other Names: Imfinzi
Drug: Tremelimumab — Dose: 300mg Route: IV

SUMMARY:
To provide early access (i.e., before marketing authorisation) to tremelimumab 300 mg IV administered once on Day 1 of Cycle 1 plus durvalumab 1500 mg IV followed by durvalumab 1500 mg IV Q4W monotherapy in patients with unresectable HCC.

DETAILED DESCRIPTION:
Overall design This is a multi centre, open-label, early access program (EAP) designed to provide treatment access to intravenous (IV) combination treatment regimen of 300 mg tremelimumab administered IV once on Day 1 of Cycle 1 plus 1500 mg durvalumab IV (MEDI 4736) followed by durvalumab IV monotherapy administered once every 4 weeks (Q4W) for eligible patients with unresectable, hepatocellular carcinoma (HCC).

Durvalumab and tremelimumab will be provided free of charge to the patients entering this program.

This global EAP will be opened in a staggered fashion, country by country, based on the requesting Treating Physician(s) and local regulations, ending when durvalumab and tremelimumab has received marketing authorisation in first line treatment in patients with unresectable hepatocellular carcinoma.

Target patient population Patients with unresectable HCC and Barcelona Clinic Liver Cancer (BCLC) stage B (who are not eligible or no longer suitable for locoregional therapy [LRT]) or stage C before entering the EAP.

Program period The EAP will enrol patients and provide resupply of durvalumab and tremelimumab until durvalumab and tremelimumab has received marketing authorisation in first line treatment for patients with unresectable HCC as per local regulations.

The EAP will be closed to new patients based on local regulations or when commercially reimbursed product is available. After reimbursement is secured, or denial of reimbursement, or decision by the Sponsor to close the enrolment, whichever occurs first, no new patients can be enrolled after this point.

In the event that market license approval or reimbursement should not be granted, contingencies will be made to ensure continued drug supply for patients who are still deriving benefit from durvalumab and tremelimumab.

Number of patients:

The number of patients who will enrol in the EAP is based on approval of unsolicited requests received from the Treating Physician.

Program treatment:

On Day 1 of Cycle 1, tremelimumab will be administered first followed by durvalumab 1 hour later. Tremelimumab will be given once on Day 1 of Cycle 1. Durvalumab monotherapy is then given Q4W.

Duration of treatment:

Patients may continue to receive EAP treatment providing they continue to show clinical benefit, as judged by the Treating Physician, in the absence of unacceptable safety concerns until disease progression, toxicity or withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over at the time of screening.
2. Body weight over 30 kg.
3. Confirmed HCC based on histopathological findings from tumour tissues.
4. Must not have received prior systemic therapy for HCC.
5. Must not be eligible for locoregional therapy for resectable HCC. For patients who progressed after locoregional therapy for HCC, locoregional therapy must have been completed at least 28 days before the baseline scan for the programme.
6. Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C (refer to Appendix H).
7. Child-Pugh Score Class A; or Child-Pugh Class B7 or B8 at discretion of treating physician (refer to Appendix I).
8. Patients with HBV infection, characterised by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV deoxyribonucleic acid (DNA) (≥10 IU/mL or above the limit of detection per local or central lab standard), must be treated with antiviral therapy, as per institutional practice to ensure adequate viral suppression (HBV DNA <2000 IU/mL) before enrolment. Patients must remain on antiviral therapy for the duration of their participation in the EAP and for 6 months after the last dose of EAP medication. Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<10 IU/mL or under the limit of detection per local or central lab standard) do not require anti-viral therapy before enrolment. These participants will be tested at every cycle to monitor HBV DNA levels and initiate anti-viral therapy if HBV DNA is detected (≥10 IU/mL or above the limit of detection per local or central lab standard). HBV DNA detectable patients must initiate and remain on anti-viral therapy for time they are in the EAP and for 6 months after the last dose of EAP medication.
9. Patients with HCV infection must have confirmed diagnosis of HCV characterised by the presence of detectable HCV ribonucleic acid (RNA) or anti-HCV antibody upon enrolment (management of this disease is per local institutional practice).
10. At least 1 measurable lesion, not previously irradiated, that can be accurately measured at baseline ≥10 mm in the longest diameter (except lymph nodes, which must have as short axis ≥15 mm) with computerised tomography (CT) or magnetic resonance imaging (MRI), and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines (Eisenhauer et al, 2009). A lesion which progressed after previous ablation or transarterial chemoembolization (TACE) could be measurable if it meets these criteria.
11. Adequate organ and marrow function, as defined below. Criteria "a", "b", "c", and "f" cannot be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose of EAP treatment.

    1. Haemoglobin ≥9 g/dL
    2. Absolute neutrophil count ≥1000/μL
    3. Platelet count ≥75,000/μL
    4. Total bilirubin (TBL) ≤2.0 x upper limit of normal (ULN)
    5. AST and ALT ≤5xULN
    6. Albumin ≥2.8 g/dL
    7. International normalised ratio (INR) ≤1.6. Note: INR prolongation due to anticoagulants for prophylaxis (e.g., atrial fibrillation) in patients without liver cirrhosis could be exception.
    8. Calculated creatinine clearance ≥50 mL/minute as determined by Cockcroft Gault (using actual body weight) or 24-hour urine creatinine clearance
12. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal as described in Section 5.3.4.
13. Must have a life expectancy of at least 12 weeks.
14. Willing and able to comply with the protocol for the duration of the EAP including undergoing treatment and scheduled visits and examination including follow up.
15. Able to provide written informed consent and any locally-required authorisation (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States [US], European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative before performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

Patients should not enter the EAP if any of the following exclusion criteria are fulfilled:

1. Concurrent enrolment in a clinical study unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study.
2. Have received an investigational product within 28 days before the first dose of EAP treatment.
3. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Grade ≥2 from previous anticancer therapy except alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Treating Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Treating Physician.
4. Any concurrent chemotherapy, study drug, or biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Known allergy or hypersensitivity to any of the EAP treatments or any of the EAP treatment excipients.
6. Child-Pugh Score Class B9; or Child-Pugh Class C
7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first dose of EAP treatments.
8. Major surgical procedure (as defined by the Treating Physician) within 28 days before the first dose of EAP treatment. Note: local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation (e.g., liver transplant).
10. History of hepatic encephalopathy within the past 12 months or requirement for medications to prevent or control encephalopathy (e.g., no lactulose, rifaximin, etc if used for purposes of hepatic encephalopathy.
11. Clinically meaningful ascites, defined as any ascites requiring non-pharmacologic intervention (e.g., paracentesis) to maintain symptomatic control, within 6 months before the first EAP treatment dose. Patients on stable doses of diuretics for ascites for ≥2 months are eligible.
12. Patients with main portal vein thrombosis (i.e., thrombosis in the main trunk of the portal vein, with or without blood flow) on baseline imaging.
13. Active or previously documented GI bleeding (e.g., oesophageal varices or ulcer bleeding) within 12 months. (Note: for patients with history of GI bleeding for >12 months or assessed as high risk for oesophageal variceal by the Treating Physician, adequate endoscopic therapy according to institutional standards is required).
14. Patient currently exhibits symptomatic or uncontrolled hypertension defined as diastolic blood pressure >90 mmHg or systolic blood pressure >140 mmHg.
15. Any condition interfering with swallowing pills, or other contraindication to oral therapy, or uncontrolled diarrhoea.
16. Active or previously documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [except for diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). Patients without active disease in the last 5 years are excluded unless discussed with the Treating Physician and considered appropriate for EAP participation. The following are exception to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients with celiac disease controlled by diet alone
17. Patients co-infected with HBV and HCV, or co-infected with HBV and hepatitis D virus (HDV). HBV positive (presence of HbsAg and/or anti-HBcAb with detectable HBV DNA); HCV positive (presence of anti-HCV antibodies); HDV positive (presence of anti-HDV antibodies).
18. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease (ILD), serious chronic GI conditions associated with diarrhoea, inferior vena cava thrombosis, or psychiatric illness/social situations that would limit compliance with EAP requirement, substantially increase the risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
19. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with known active disease ≥5 years before the first dose of EAP treatment and of low potential risk for recurrence
    * Patients with a history of prostate cancer of stage <T2cN0M0 without biochemical recurrence or progression and who, in the opinion of the Treating Physician are not deemed to require active intervention
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
20. History of leptomeningeal carcinomatosis.
21. History of, or current, brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT, each preferably with IV contrast of the brain before EAP entry.
22. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
23. History of active primary immunodeficiency.
24. Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), or human immunodeficiency virus (HIV; positive HIV 1/2 antibodies).
25. Current or prior use of immunosuppressive medication within 14 days before the first dose of EAP treatment. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as pre-medication for hypersensitivity reactions (e.g., CT scan pre-medication)
26. Receipt of live attenuated vaccine within 30 days before the first dose of EAP treatment. Note: patients, if enrolled, should not receive live vaccine while receiving EAP treatments, and up to 30 days after the last dose of EAP treatment.
27. Female patients who are pregnant or breastfeeding, or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab+tremelimumab or 90 days after the last dose of durvalumab monotherapy. Not engaging in sexual activity, as per the patient's preferred and usual lifestyle, for the total duration of the treatment and washout periods is an acceptable practice.
28. Previous randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
29. Patients who have received anti-PD-1, anti-PD-L1, or anti-CTLA-4 before the first dose of EAP treatment.
30. Patient has any condition that, in the opinion of the Treating Physician would interfere with the evaluation of the programme drug or interpretation of patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Newark, Delaware
  - Research Site, Minneapolis, Minnesota
  - Research Site, Reno, Nevada
  - Research Site, Morgantown, West Virginia